CLINICAL TRIAL: NCT04543643
Title: Endoscopic and Microbiological Assessment of the Effect of Carvedilol Combined With Berberine on GOV in Cirrhosis: a Prospective Cohort Study
Brief Title: Endoscopic and Microbiological Assessment of the Effect of Carvedilol Combined With Berberine on GOV in Cirrhosis
Acronym: CABER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tianjin2PH
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Cirrhosis Due to Hepatitis B; Cirrhosis Due to Hepatitis C; Gastroesophageal Varices
Keywords: gastroesophageal varices; cirrhosis; carvedilol; berberine; Endoscopic ultrasonography; gut microbiota; portal hypertension
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Carvedilol; Berberine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carvedilol+ berberine (Experimental): Carvedilol is started at a dose of 6.25 mg once per day. After 1 week, this will increased to a dose of 6.25 mg twice daily per day if systolic blood pressure does not fall below 85mm Hg and HR 55/min. Berberine is started at a dose of 0.3g twice per day.
  Interventions: Drug: Carvedilol; Drug: Berberine
- Carvedilol (Active Comparator): Carvedilol is started at a dose of 6.25 mg once per day. After 1 week, this will increased to a dose of 6.25 mg twice daily per day if systolic blood pressure does not fall below 85 mm Hg and HR 55/min.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — As the third generation of NSBB, carvedilol is more effective in reducing HVPG than propranolol, which is recommended by Baveno VI as the first-line drug for EVB primary prevention.
Drug: Berberine — Berberine can regulate the intestinal flora, which is safe and effective in clinical application.
  Arms: Carvedilol+ berberine

SUMMARY:
Carvedilol has been shown to be more potent in decreasing portal hypertension to propranolol. A lot of studies have shown that the imbalance of flora and the progress of portal hypertension are mutually causal. Berberine can regulate the intestinal flora.In this study, we evaluated the effect of carvedilol and berberine on reducing portal vein pressure by observing the changes of endoscopy，endoscopic ultrasonography and intestinal flora.

DETAILED DESCRIPTION:
There is a higher risk of esophageal and gastric varices bleeding in cirrhosis patients with moderate and severe esophageal and gastric varices. Once there is a high mortality rate of esophageal and gastric varices bleeding, it will cause great losses to the family and society. Therefore, it is of great social and economic significance to prevent esophageal and gastric varices bleeding through economic and effective methods. As the third generation of NSBB, carvedilol is more effective in reducing HVPG than propranolol, which is recommended by Baveno VI as the first-line drug for EVB primary prevention. A lot of studies have shown that the imbalance of flora and the progress of portal hypertension are mutually causal. The application of carvedilol can reduce the pressure of portal vein, and when the portal hypertension is improved, the imbalance of intestinal mucosal barrier and flora will also be changed. Berberine can regulate the intestinal flora, which is safe and effective in clinical application. Gastroscopy is still the main method of screening varicose veins. We can determine whether there is GOV in patients and evaluate the risk of varicose vein bleeding. However, gastroscopy can only observe the situation in the digestive tract lumen, and ultrasound endoscopy can scan the outside of the tube wall, so as to more comprehensively evaluate the change of portal hypertension. The purpose of this study is to apply endoscopic ultrasonography to the whole process of the study, which can be used as a more sensitive means to observe the changes of portal hypertension, and to systematically evaluate the continuous changes of portal hypertension. It provides a theoretical basis and measurement means for a more comprehensive and scientific evaluation of portal hypertension.In this study, the patients with GOV who need primary prevention were randomly divided into two groups. Carvedilol or carvedilol combined with berberine were given for 12 months respectively. The degree of varicose vein relief was judged by ES and EUS, and the changes of oral and intestinal flora were detected at the same time To understand the possible mechanism of carvedilol and berberine in reducing portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* HBV-related or/and HCV-related liver cirrhotic patients based on pathology or clinical diagnosis;

  * Antiviral therapy;
  * Male or Female;
  * ES showed the presence of esophageal and gastric varices and / or red signs;
  * Child-Pugh < 10, and meld < 29;
  * Signature of informed consent.

Exclusion Criteria:

* • Used antibiotics, prebiotics, probiotics and proton pump inhibitors within 2 weeks;

  * Any contra-indications to beta-blockers including asthma, chronic obstructive pulmonary disease, allergic rhinitis, NYHA (New York Heart Association) class IV heart failure, atrioventricular block, sinus bradycardia (HR < 50 / min), cardiogenic shock, hypotension (SBP < 85mmHg), sick sinus syndrome, insulin dependent diabetes, peripheral vascular disease;
  * Unstable high blood pressure and long-term engagement in driving;
  * Any malignancy that affects survival, excluding the cured;
  * Patients with portal thrombosis;
  * PT extension greater than 4 seconds, PLT<30×10^9/L;
  * Pregnant and lactating patients;
  * History of surgery for portal hypertension；History of prior EVL (endoscopic variceal ligation) or sclerotherapy, history of surgery for portal hypertension including portosystemic shunts, disconnection and spleen resection and transjugular intrahepatic portosystemic shunt;
  * Patients with severe diseases of vital organs such as heart, lung, kidney, brain, blood and nervous system;
  * Allergic to carvedilol and berberine;
  * Severe systemic diseases；
  * hemolytic anemia and lack of glucose - 6 - phosphate dehydrogenase patients
  * Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
The progression Incidence of esophageal varices | 1 year
  progression of esophagogastric varices under gastroscopy and/or endoscopic ultrasound

SECONDARY OUTCOMES:
The incidence of liver cirrhosis decompensation | 1 year
  the occurrence of decompensating events in cirrhosis (decompensating is defined as gastrointestinal bleeding, ascites, or significant hepatic encephalopathy, hepatorenal syndrome, associated with portal hypertension)
HCC, death or liver transplantation | 1 year
  The incidence of hepatic cellular carcinoma, death or liver transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Second People's Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Result] North Italian Endoscopic Club for the Study and Treatment of Esophageal Varices. Prediction of the first variceal hemorrhage in patients with cirrhosis of the liver and esophageal varices. A prospective multicenter study. N Engl J Med. 1988 Oct 13;319(15):983-9. doi: 10.1056/NEJM198810133191505. PMID 3262200
- [Result] Carbonell N, Pauwels A, Serfaty L, Fourdan O, Levy VG, Poupon R. Improved survival after variceal bleeding in patients with cirrhosis over the past two decades. Hepatology. 2004 Sep;40(3):652-9. doi: 10.1002/hep.20339. PMID 15349904
- [Result] Wang X, Lin SX, Tao J, Wei XQ, Liu YT, Chen YM, Wu B. Study of liver cirrhosis over ten consecutive years in Southern China. World J Gastroenterol. 2014 Oct 7;20(37):13546-55. doi: 10.3748/wjg.v20.i37.13546. PMID 25309085
- [Result] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Result] Abadia M, Montes ML, Ponce D, Froilan C, Romero M, Poza J, Hernandez T, Fernandez-Martos R, Olveira A; "La Paz Portal Hypertension" Study Group Investigators. Management of betablocked patients after sustained virological response in hepatitis C cirrhosis. World J Gastroenterol. 2019 Jun 7;25(21):2665-2674. doi: 10.3748/wjg.v25.i21.2665. PMID 31210717
- [Result] Hammoud GM, Ibdah JA. Utility of endoscopic ultrasound in patients with portal hypertension. World J Gastroenterol. 2014 Oct 21;20(39):14230-6. doi: 10.3748/wjg.v20.i39.14230. PMID 25339809
- [Result] Hashizume M, Kitano S, Sugimachi K, Sueishi K. Three-dimensional view of the vascular structure of the lower esophagus in clinical portal hypertension. Hepatology. 1988 Nov-Dec;8(6):1482-7. doi: 10.1002/hep.1840080603. PMID 3192160
- [Result] Huang JY, Samarasena JB, Tsujino T, Chang KJ. EUS-guided portal pressure gradient measurement with a novel 25-gauge needle device versus standard transjugular approach: a comparison animal study. Gastrointest Endosc. 2016 Aug;84(2):358-62. doi: 10.1016/j.gie.2016.02.032. Epub 2016 Mar 3. PMID 26945557
- [Result] Tripathi D, Ferguson JW, Kochar N, Leithead JA, Therapondos G, McAvoy NC, Stanley AJ, Forrest EH, Hislop WS, Mills PR, Hayes PC. Randomized controlled trial of carvedilol versus variceal band ligation for the prevention of the first variceal bleed. Hepatology. 2009 Sep;50(3):825-33. doi: 10.1002/hep.23045. PMID 19610055
- [Result] Reiberger T, Ulbrich G, Ferlitsch A, Payer BA, Schwabl P, Pinter M, Heinisch BB, Trauner M, Kramer L, Peck-Radosavljevic M; Vienna Hepatic Hemodynamic Lab. Carvedilol for primary prophylaxis of variceal bleeding in cirrhotic patients with haemodynamic non-response to propranolol. Gut. 2013 Nov;62(11):1634-41. doi: 10.1136/gutjnl-2012-304038. Epub 2012 Dec 18. PMID 23250049
- [Result] Bhardwaj A, Kedarisetty CK, Vashishtha C, Bhadoria AS, Jindal A, Kumar G, Choudhary A, Shasthry SM, Maiwall R, Kumar M, Bhatia V, Sarin SK. Carvedilol delays the progression of small oesophageal varices in patients with cirrhosis: a randomised placebo-controlled trial. Gut. 2017 Oct;66(10):1838-1843. doi: 10.1136/gutjnl-2016-311735. Epub 2016 Jun 13. PMID 27298379
- [Result] Borzio M, Salerno F, Piantoni L, Cazzaniga M, Angeli P, Bissoli F, Boccia S, Colloredo-Mels G, Corigliano P, Fornaciari G, Marenco G, Pistara R, Salvagnini M, Sangiovanni A. Bacterial infection in patients with advanced cirrhosis: a multicentre prospective study. Dig Liver Dis. 2001 Jan-Feb;33(1):41-8. doi: 10.1016/s1590-8658(01)80134-1. PMID 11303974
- [Result] Pascual S, Such J, Esteban A, Zapater P, Casellas JA, Aparicio JR, Girona E, Gutierrez A, Carnices F, Palazon JM, Sola-Vera J, Perez-Mateo M. Intestinal permeability is increased in patients with advanced cirrhosis. Hepatogastroenterology. 2003 Sep-Oct;50(53):1482-6. PMID 14571769
- [Result] Garcia-Tsao G. Bacterial translocation: cause or consequence of decompensation in cirrhosis? J Hepatol. 2001 Jan;34(1):150-5. doi: 10.1016/s0168-8278(00)00006-4. No abstract available. PMID 11211893
- [Result] Arvaniti V, D'Amico G, Fede G, Manousou P, Tsochatzis E, Pleguezuelo M, Burroughs AK. Infections in patients with cirrhosis increase mortality four-fold and should be used in determining prognosis. Gastroenterology. 2010 Oct;139(4):1246-56, 1256.e1-5. doi: 10.1053/j.gastro.2010.06.019. Epub 2010 Jun 14. PMID 20558165
- [Result] Goulis J, Armonis A, Patch D, Sabin C, Greenslade L, Burroughs AK. Bacterial infection is independently associated with failure to control bleeding in cirrhotic patients with gastrointestinal hemorrhage. Hepatology. 1998 May;27(5):1207-12. doi: 10.1002/hep.510270504. PMID 9581672
- [Result] Thalheimer U, Triantos CK, Samonakis DN, Patch D, Burroughs AK. Infection, coagulation, and variceal bleeding in cirrhosis. Gut. 2005 Apr;54(4):556-63. doi: 10.1136/gut.2004.048181. No abstract available. PMID 15753544
- [Result] Reiberger T, Ferlitsch A, Payer BA, Mandorfer M, Heinisch BB, Hayden H, Lammert F, Trauner M, Peck-Radosavljevic M, Vogelsang H; Vienna Hepatic Hemodynamic Lab. Non-selective betablocker therapy decreases intestinal permeability and serum levels of LBP and IL-6 in patients with cirrhosis. J Hepatol. 2013 May;58(5):911-21. doi: 10.1016/j.jhep.2012.12.011. Epub 2012 Dec 20. PMID 23262249
- [Result] Adamberg K, Tomson K, Talve T, Pudova K, Puurand M, Visnapuu T, Alamae T, Adamberg S. Levan Enhances Associated Growth of Bacteroides, Escherichia, Streptococcus and Faecalibacterium in Fecal Microbiota. PLoS One. 2015 Dec 2;10(12):e0144042. doi: 10.1371/journal.pone.0144042. eCollection 2015. PMID 26629816
- [Result] Yao J, Chang L, Yuan L, Duan Z. Nutrition status and small intestinal bacterial overgrowth in patients with virus-related cirrhosis. Asia Pac J Clin Nutr. 2016;25(2):283-91. doi: 10.6133/apjcn.2016.25.2.06. PMID 27222411
- [Result] Hoyles L, Fernandez-Real JM, Federici M, Serino M, Abbott J, Charpentier J, Heymes C, Luque JL, Anthony E, Barton RH, Chilloux J, Myridakis A, Martinez-Gili L, Moreno-Navarrete JM, Benhamed F, Azalbert V, Blasco-Baque V, Puig J, Xifra G, Ricart W, Tomlinson C, Woodbridge M, Cardellini M, Davato F, Cardolini I, Porzio O, Gentileschi P, Lopez F, Foufelle F, Butcher SA, Holmes E, Nicholson JK, Postic C, Burcelin R, Dumas ME. Molecular phenomics and metagenomics of hepatic steatosis in non-diabetic obese women. Nat Med. 2018 Jul;24(7):1070-1080. doi: 10.1038/s41591-018-0061-3. Epub 2018 Jun 25. PMID 29942096
- [Result] Silva Santos PS, Fernandes KS, Gallottini MH. Assessment and management of oral health in liver transplant candidates. J Appl Oral Sci. 2012 Mar-Apr;20(2):241-5. doi: 10.1590/s1678-77572012000200020. PMID 22666844
- [Result] Aberg F, Helenius-Hietala J, Meurman J, Isoniemi H. Association between dental infections and the clinical course of chronic liver disease. Hepatol Res. 2014 Mar;44(3):349-53. doi: 10.1111/hepr.12126. Epub 2013 Apr 29. PMID 23607641
- [Result] Bajaj JS, Betrapally NS, Hylemon PB, Heuman DM, Daita K, White MB, Unser A, Thacker LR, Sanyal AJ, Kang DJ, Sikaroodi M, Gillevet PM. Salivary microbiota reflects changes in gut microbiota in cirrhosis with hepatic encephalopathy. Hepatology. 2015 Oct;62(4):1260-71. doi: 10.1002/hep.27819. Epub 2015 May 6. PMID 25820757
- [Result] Wang Y, Shou JW, Li XY, Zhao ZX, Fu J, He CY, Feng R, Ma C, Wen BY, Guo F, Yang XY, Han YX, Wang LL, Tong Q, You XF, Lin Y, Kong WJ, Si SY, Jiang JD. Berberine-induced bioactive metabolites of the gut microbiota improve energy metabolism. Metabolism. 2017 May;70:72-84. doi: 10.1016/j.metabol.2017.02.003. Epub 2017 Feb 10. PMID 28403947
- [Result] Chen YX, Gao QY, Zou TH, Wang BM, Liu SD, Sheng JQ, Ren JL, Zou XP, Liu ZJ, Song YY, Xiao B, Sun XM, Dou XT, Cao HL, Yang XN, Li N, Kang Q, Zhu W, Xu HZ, Chen HM, Cao XC, Fang JY. Berberine versus placebo for the prevention of recurrence of colorectal adenoma: a multicentre, double-blinded, randomised controlled study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):267-275. doi: 10.1016/S2468-1253(19)30409-1. Epub 2020 Jan 8. PMID 31926918
- [Result] Mandorfer M, Peck-Radosavljevic M, Reiberger T. Prevention of progression from small to large varices: are we there yet? An updated meta-analysis. Gut. 2017 Jul;66(7):1347-1349. doi: 10.1136/gutjnl-2016-312814. Epub 2016 Sep 30. No abstract available. PMID 27694143
- [Result] Sharma M, Singh S, Desai V, Shah VH, Kamath PS, Murad MH, Simonetto DA. Comparison of Therapies for Primary Prevention of Esophageal Variceal Bleeding: A Systematic Review and Network Meta-analysis. Hepatology. 2019 Apr;69(4):1657-1675. doi: 10.1002/hep.30220. Epub 2019 Feb 20. PMID 30125369
- [Result] Shah HA, Azam Z, Rauf J, Abid S, Hamid S, Jafri W, Khalid A, Ismail FW, Parkash O, Subhan A, Munir SM. Carvedilol vs. esophageal variceal band ligation in the primary prophylaxis of variceal hemorrhage: a multicentre randomized controlled trial. J Hepatol. 2014 Apr;60(4):757-64. doi: 10.1016/j.jhep.2013.11.019. Epub 2013 Nov 28. PMID 24291366
- [Result] Schwarzer R, Kivaranovic D, Paternostro R, Mandorfer M, Reiberger T, Trauner M, Peck-Radosavljevic M, Ferlitsch A. Carvedilol for reducing portal pressure in primary prophylaxis of variceal bleeding: a dose-response study. Aliment Pharmacol Ther. 2018 Apr;47(8):1162-1169. doi: 10.1111/apt.14576. Epub 2018 Feb 28. PMID 29492989
- [Result] Ding Q, Tian XG, Li Y, Wang QZ, Zhang CQ. Carvedilol may attenuate liver cirrhosis by inhibiting angiogenesis through the VEGF-Src-ERK signaling pathway. World J Gastroenterol. 2015 Aug 28;21(32):9566-76. doi: 10.3748/wjg.v21.i32.9566. PMID 26327764
- [Result] Gupta N, Kumar A, Sharma P, Garg V, Sharma BC, Sarin SK. Effects of the adjunctive probiotic VSL#3 on portal haemodynamics in patients with cirrhosis and large varices: a randomized trial. Liver Int. 2013 Sep;33(8):1148-57. doi: 10.1111/liv.12172. Epub 2013 Apr 21. PMID 23601333
- [Result] Kakiyama G, Pandak WM, Gillevet PM, Hylemon PB, Heuman DM, Daita K, Takei H, Muto A, Nittono H, Ridlon JM, White MB, Noble NA, Monteith P, Fuchs M, Thacker LR, Sikaroodi M, Bajaj JS. Modulation of the fecal bile acid profile by gut microbiota in cirrhosis. J Hepatol. 2013 May;58(5):949-55. doi: 10.1016/j.jhep.2013.01.003. Epub 2013 Jan 16. PMID 23333527
- [Result] Szabo G. Gut-liver axis in alcoholic liver disease. Gastroenterology. 2015 Jan;148(1):30-6. doi: 10.1053/j.gastro.2014.10.042. Epub 2014 Nov 11. PMID 25447847
- [Result] Seo YS, Shah VH. The role of gut-liver axis in the pathogenesis of liver cirrhosis and portal hypertension. Clin Mol Hepatol. 2012 Dec;18(4):337-46. doi: 10.3350/cmh.2012.18.4.337. Epub 2012 Dec 21. PMID 23323248
- [Result] Bernardi M, Moreau R, Angeli P, Schnabl B, Arroyo V. Mechanisms of decompensation and organ failure in cirrhosis: From peripheral arterial vasodilation to systemic inflammation hypothesis. J Hepatol. 2015 Nov;63(5):1272-84. doi: 10.1016/j.jhep.2015.07.004. Epub 2015 Jul 17. PMID 26192220
- [Result] Moghadamrad S, McCoy KD, Geuking MB, Sagesser H, Kirundi J, Macpherson AJ, De Gottardi A. Attenuated portal hypertension in germ-free mice: Function of bacterial flora on the development of mesenteric lymphatic and blood vessels. Hepatology. 2015 May;61(5):1685-95. doi: 10.1002/hep.27698. Epub 2015 Feb 24. PMID 25643846
- [Result] Garcia-Lezana T, Raurell I, Bravo M, Torres-Arauz M, Salcedo MT, Santiago A, Schoenenberger A, Manichanh C, Genesca J, Martell M, Augustin S. Restoration of a healthy intestinal microbiota normalizes portal hypertension in a rat model of nonalcoholic steatohepatitis. Hepatology. 2018 Apr;67(4):1485-1498. doi: 10.1002/hep.29646. Epub 2018 Feb 19. PMID 29113028
- [Result] European Association for the Study of the Liver. EASL Recommendations on Treatment of Hepatitis C 2018. J Hepatol. 2018 Aug;69(2):461-511. doi: 10.1016/j.jhep.2018.03.026. Epub 2018 Apr 9. No abstract available. PMID 29650333
- [Result] Feng R, Shou JW, Zhao ZX, He CY, Ma C, Huang M, Fu J, Tan XS, Li XY, Wen BY, Chen X, Yang XY, Ren G, Lin Y, Chen Y, You XF, Wang Y, Jiang JD. Transforming berberine into its intestine-absorbable form by the gut microbiota. Sci Rep. 2015 Jul 15;5:12155. doi: 10.1038/srep12155. PMID 26174047
- [Result] Koren O, Goodrich JK, Cullender TC, Spor A, Laitinen K, Backhed HK, Gonzalez A, Werner JJ, Angenent LT, Knight R, Backhed F, Isolauri E, Salminen S, Ley RE. Host remodeling of the gut microbiome and metabolic changes during pregnancy. Cell. 2012 Aug 3;150(3):470-80. doi: 10.1016/j.cell.2012.07.008. PMID 22863002